CLINICAL TRIAL: NCT02397551
Title: Supplementing the Luteal Phase With Three Small Doses of HCG Versus Booster Dose of HCG on Ovum Pickup Day in Antagonist IVF/ICSI Cycles Triggered With GnRH Agonist in High Responder Females to Salvage the Luteal Phase
Brief Title: Three Small Doses of HCG Versus Booster Dose of HCG on Ovum Pickup Day
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Nile Ivf Center, Cairo, Egypt (Other); Adam International Hospital (Other)
Responsible Party: Principal Investigator, Yasmin Ahmed Bassiouny, Dr, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22015
Record Dates: First submitted 2015-03-16; First posted 2015-03-25 (Estimated); Last update posted 2018-01-29 (Actual); Status verified 2018-01

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Chorionic Gonadotropin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Small doses of HCG (Active Comparator): Supplementing the luteal phase with three small doses (500 IU) of HCG after trigger with GnRH agonist in antagonist IVF/ICSI cycles in high responders
  Interventions: Procedure: IVF/ICSI; Drug: Human Chorionic Gonadotropin
- Booster HCG dose (Active Comparator): Booster HCG dose GnRH agonist only to trigger final maturation followed by a booster dose of 1500 IU of HCG on the day of ovum pickup
  Interventions: Procedure: IVF/ICSI; Drug: Human Chorionic Gonadotropin

INTERVENTIONS:
Procedure: IVF/ICSI
Drug: Human Chorionic Gonadotropin — Given in different doses and timing to support the luteal phase

SUMMARY:
To salvage the luteal phase and improve pregnancy rate in antagonist IVF/ICSI cycles triggered with GnRH agonist. Two strategies are compared supplementing the luteal phase with three small doses (500 IU) of HCG and giving a booster dose of HCG (1500 IU) on the day of ovum pickup.

ELIGIBILITY:
Inclusion Criteria:

* High responder females undergoing antagonist protocol IVF/ICSI cycle
* More than 14 MII oocytes
* Estradiol more than 3500 pg/ml on day of trigger

Exclusion Criteria:

* Any other protocol
* Normal or poor responders

Ages: 20 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy rate | 1 year
  The number of cycles with a positive pregnancy test and evidence of a gestational sac with fetal pulsations after 5weeks from pregnancy test

SECONDARY OUTCOMES:
OHSS rate | 1 year
  The number of cycles with evidence of OHSS

OTHER OUTCOMES:
Chemical pregnancy rate | 1 year
  The number of cycles with a positive pregnancy test after 14 days from embryo transfer
Early miscarriage rate | 1 year
  Pregnancies that end up with miscarriage before 12 weeks gestation
Ongoing pregnancy rate | 1 year
  Pregnancies ongoing beyond 12 weeks gestation
Live birth rate | 1 year
  Pregnancies resulting in a live birth

CONTACTS AND LOCATIONS:
Overall Officials: Sarwat Ahwany, MD, Study Director — Cairo University
Locations (3):
- Egypt (3):
  - IVF centre, Obstetrics and Gynaecology Department, Cairo University Hospitals (Kasr EL Aini), Cairo
  - Adam International hospital, Giza
  - Nile IVF center, Giza